CLINICAL TRIAL: NCT02376114
Title: The Effect of Ginkgo Biloba on Ocular Blood Flow in Primary Open-Angle Glaucoma Patients: A Double-Blind Randomized Crossover Trial
Brief Title: Ginkgo Biloba and Ocular Blood Flow in Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Ellen Freeman, Associate Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ginkgo and blood flow
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma, Open-Angle
Keywords: ocular blood flow; ginkgo biloba; glaucoma; vasospasm
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ginkgo-Placebo (Other): Patients receive Ginkgo biloba and then placebo afterwards.
  Interventions: Drug: Ginkgo biloba
- Placebo-Ginkgo (Other): Patients receive placebo and then Ginkgo biloba afterwards.
  Interventions: Drug: Placebo to Ginkgo biloba

INTERVENTIONS:
Drug: Ginkgo biloba — The Ginkgo biloba extract that was used contained 24% ginkgo flavone glycosides and 6% terpene lactones (Vitamin Research Products, Carson City, Nevada). Patients took 60 mg of Ginkgo or a placebo twice daily by mouth for two weeks. The placebo consisted of 40 mg of corn starch. Ginkgo and the placebo were encapsulated to ensure identical appearance.
  Arms: Ginkgo-Placebo
Drug: Placebo to Ginkgo biloba
  Arms: Placebo-Ginkgo

SUMMARY:
Glaucoma is one of the leading causes of blindness. Ginkgo biloba may be part of an effective treatment strategy for glaucoma because it has been shown to improve blood flow, it has antioxidant properties, it can relax smooth muscle, and it can protect neurons from damage. The goal of our study was to determine whether Ginkgo biloba would result in increased ocular blood flow which may protect against glaucoma damage.

DETAILED DESCRIPTION:
Glaucoma is one of the leading causes of blindness. Glaucoma progression sometimes occurs despite apparent control of intraocular pressure. Therefore, there may be other factors involved in glaucoma progression in some patients. Evidence is mounting that glaucoma patients are more likely to have abnormal ocular blood flow and vasospasm compared to those without glaucoma. Also, a study showed that those with progressive glaucoma had decreased blood flow compared to those with stable glaucoma or healthy controls. Endothelin-1, a potent vasoconstrictor, may be involved in these blood flow abnormalities. If the dysregulation of blood flow is causally related to the progression of glaucoma, then therapies aimed at improving the regulation of blood flow may help to prevent this progression.

Ginkgo may be part of an effective treatment strategy for glaucoma because it has been shown to improve peripheral and cerebral blood flow. Other properties of Ginkgo that may aid in the treatment of glaucoma include antioxidant properties, inhibition of platelet activating factor, relaxation of smooth muscle, and neuroprotective properties. Ginkgo may be particularly useful in relaxing vasospasm. Two controlled trials have examined the effect of Ginkgo on ocular blood flow in healthy subjects. One randomized crossover trial found that 2 days of Ginkgo increased the end diastolic velocity in the ophthalmic artery compared to placebo. However, another trial found that 1 dose of Ginkgo had no significant effects on ocular blood flow parameters. In people with normal tension glaucoma, Park et al found that 4 weeks of Ginkgo increased peripapillary retinal blood flow. Two randomized controlled trials have examined the impact of Ginkgo biloba on visual field in people with normal tension glaucoma with conflicting results. Clearly, there is a need for more research on this topic.

The goal of our study was to determine whether Ginkgo biloba would result in increased ocular blood flow, reduced vasospasm, and reduced endothelin-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* We focused this trial on vasospastic glaucoma patients because we believed that these would be the patients most likely to benefit from the ability of Ginkgo to improve blood flow.
* Patients who had been identified from previous research as being vasospastic on the Transonic Laser Doppler Flowmeter (Transonic Systems Inc., Ithaca, NY) were contacted and asked if they would like to participate in the trial.
* We recruited vasospastic patients with early or moderate primary open-angle glaucoma with a typical visual field defect with an abnormal Glaucoma Hemifield Test and a Mean Deviation worse than -2 decibels, and an optic nerve head showing retinal nerve fiber layer or neuroretinal rim loss characteristic of glaucoma.
* There was no restriction for intraocular pressure at time of diagnosis although at the time of recruitment intraocular pressure had to be effectively controlled either by ocular hypertension therapy or by surgery.
* If a patient had two eyes eligible, data from the right eye only was used.

Exclusion Criteria:

* those taking anticoagulant therapy,
* those with blood disorders or diabetes,
* women who were pregnant, planning to become pregnant, or who were breast-feeding,
* patients with a history of seizures or who were currently taking anti-convulsant medication, and
* those who could not return for 2 follow-up visits at 4 and 6 weeks.
* those patients who are already taking Ginkgo were asked if they were willing to stop for 6 weeks before the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in optic nerve head blood flow in the rim region as measured with the Heidelberg Retinal Flowmeter | 4 weeks and 10 weeks
  Change in optic nerve head blood flow in the rim region as measured with the Heidelberg Retinal Flowmeter

SECONDARY OUTCOMES:
Change in retinal blood flow as measured by the Canon Laser Blood Flowmeter | 4 weeks and 10 weeks
  Change in retinal blood flow as measured by the Canon Laser Blood Flowmeter
Change in ocular pulse amplitude as measured with the Pascal Dynamic Contour Tonometer | 4 weeks and 10 weeks
  Change in ocular pulse amplitude as measured with the Pascal Dynamic Contour Tonometer
Change in peripheral vasospasm as measured during the cold provocation test using the Transonic Laser Doppler Flowmeter | 4 weeks and 10 weeks
  Change in peripheral vasospasm as measured during the cold provocation test as measured using the Transonic Laser Doppler Flowmeter
Change in endothelin-1 levels as measured by an enzyme-linked immunosorbent assay kit | 4 weeks and 10 weeks
  Change in endothelin-1 levels as measured by an enzyme-linked immunosorbent assay kit

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Freeman, PhD, Principal Investigator — Maisonneuve-Rosemont Hospital; Mark Lesk, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada